CLINICAL TRIAL: NCT05065671
Title: Incorporating Drug Metabolism by the Human Gut Microbiome Into Personalized Medicine
Brief Title: Microbiome Derived Metabolism and Pharmacokinetics
Acronym: MDM-PK
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Luigi Brunetti, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro2021000945
Record Dates: First submitted 2021-09-13; First posted 2021-10-04 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-03

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Tolcapone; Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tolcapone (Experimental): Tolcapone 100 mg by mouth once
  Interventions: Drug: Tolcapone 100 MG
- Duloxetine (Experimental): Duloxetine 20 mg by mouth once
  Interventions: Drug: Duloxetine 20 MG

INTERVENTIONS:
Drug: Tolcapone 100 MG — Tolcapone 100 mg by mouth once
  Arms: Tolcapone
Drug: Duloxetine 20 MG — Duloxetine 20 mg by mouth once
  Arms: Duloxetine

SUMMARY:
The investigators will perform single-dose pharmacokinetic (PK) studies in humans following administration of drugs with known microbiome derived metabolism (MDM) in parallel with preclinical studies. By directly comparing laboratory measurements to clinical results, the investigators will be able to confirm the relevance of MDM in vivo, create microbiome-dependent PK profiles of the MDM positive drugs, and establish methodology to capture the contribution of MDM to inter-individual variability in clinical drug PK profiles.

DETAILED DESCRIPTION:
The human gut microbiome has been shown to play an important role in the observed inter-individual variability in therapeutic response, including both efficacy and toxicity. One of the mechanisms by which the gut microbiome exerts these effects is through the direct biochemical transformation of orally administered drugs into more or less active or toxic metabolites, termed herein microbiome-derived drug metabolism (MDM). Recent systematic studies have revealed an enormous and largely unexplored biochemical capacity of human gut bacteria - cultured in ex vivo microbial communities or as single isolates - to metabolize dozens of orally administered drugs but the clinical relevance of the observed MDM remains unmapped. This gap in knowledge is a result of overt disconnect between preclinical and clinical studies: MDM studies performed in the laboratory are removed from direct clinical comparisons, and human studies performed during drug development and therapeutic interventions almost completely ignore microbiome contribution. Moreover, there is currently a lack standardized experimental methods and mathematical models to start incorporating MDM into clinical decisions. Our PK studies are aimed at developing such strategies into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Body mass index between 18.5 - 29.9 kg/m2

Exclusion Criteria

* Estimated creatinine clearance < 50 mL/min
* Liver impairment (liver enzymes > 2 times upper limit)
* Antibiotics in the past 3 months
* History of gastrointestinal disease
* History of autoimmune disorder
* Chronic viral infection
* Smoker
* Alcohol intake (defined as having up to 1 drink per day for women and up to 2 drinks per day for men)
* Use of immune modulating medications
* Diabetes mellitus
* Any history or contraindication to the study medications
* Additional exclusion criteria will be based on the FDA approved prescribing information for selected drugs (i.e., contraindications)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Drug area under the plasma concentration versus time curve (AUC) | After a single dose of a microbiome derived metabolism positive drug (over an 8 hour period for each drug)
  We will calculate the plasma area under the curve for the microbiome derived metabolism positive probe drugs
Drug peak plasma concentration | After a single dose of a microbiome derived metabolism positive drug (over an 8 hour period for each drug)
  We will measure the peak plasma concentration for microbiome derived metabolism positive probe drugs
Drug trough plasma concentrations | After a single dose of a microbiome derived metabolism positive drug (over an 8 hour period for each drug)
  We will measure the trough plasma concentration for microbiome derived metabolism positive probe drugs
Drug volume of distribution | After a single dose of a microbiome derived metabolism positive drug (over an 8 hour period for each drug)
  We will calculate the volume of distribution for microbiome derived metabolism positive probe drugs
Drug half-life | After a single dose of a microbiome derived metabolism positive drug (over an 8 hour period for each drug)
  We will calculate drug half-life for microbiome derived metabolism positive probe drugs
Drug plasma clearance | After a single dose of a microbiome derived metabolism positive drug (over an 8 hour period for each drug)
  We will calculate drug plasma clearance for each microbiome derived metabolism positive drug.

OTHER OUTCOMES:
Quantitation of microbiome derived metabolism positive drug metabolites in urine | After a single dose of a microbiome derived metabolism positive drug (over an 8 hour period for each drug)
  The concentration of microbiome derived metabolism positive drug metabolites in urine will be measured
Quantitation of microbiome derived metabolism positive drugs in urine | After a single dose of a microbiome derived metabolism positive drug (over an 8 hour period for each drug)
  The concentration of microbiome derived metabolism positive drugs in urine will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No